CLINICAL TRIAL: NCT06186674
Title: Prediction of Back Disability Using Clinical, Functional, and Bio-mechanical Variables in Adults With Low Back Pain
Brief Title: Prediction of Back Disability in Adults With Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Aliaa Mohamed Elabd, lecturer, basic science department, faculty of physical therapy, benha university, Benha University
Other Study IDs: PT.BU.EC.1
Record Dates: First submitted 2023-12-07; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
Keywords: posture
MeSH Terms: conditions — Low Back Pain | interventions — Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal: normal persons
  Interventions: Diagnostic Test: sorensen test for back endurance; Diagnostic Test: 6 minute walk test; Diagnostic Test: c7-s1 SVA
- low back pain: patients with low back pain
  Interventions: Diagnostic Test: sorensen test for back endurance; Diagnostic Test: 6 minute walk test; Diagnostic Test: c7-s1 SVA

INTERVENTIONS:
Diagnostic Test: sorensen test for back endurance — • Biering-Sorensen test will be utilized to gauge the trunk extensor muscles' isometric endurance. The patient will be lying on a treatment couch, prone. The top half of the body will be permitted to rest on a chair prior to the test starting. The patient will be told to elevate their upper trunks off of the chair at the start of the test. the examiner determined how long the individual could hold this position.
Diagnostic Test: 6 minute walk test — It gauges how far a person can go while walking for a total of six minutes on a level, hard surface. Cones will be used to mark turns at the start and end of the 30-meter border and every three meters throughout the corridor or walkway that was utilized for the test. The patient's objective is to cover the most distance in six minutes at a reasonable pace.
  It gauges how far a person can go while walking for a total of six minutes on a level, hard surface. Cones will be used to mark turns at the start and end of the 30-meter border and every three meters throughout the corridor or walkway that was utilized for the test. The patient's objective is to cover the most distance in six minutes at a reasonable pace.
Diagnostic Test: c7-s1 SVA — Subjects will obtain standardized lateral views radiographs in a neutral standing position for the whole spine. The C7- S1 SVA will be measured as the distance from the plumb line dropped from the center of the C7 vertebral body to the most posterior edge of the upper sacral endplate surface.

SUMMARY:
Low back pain (LBP) is one of the most enormous and challenging disorders. LBP represents a leading cause of disability worldwide. A number of variables (clinical, functional and mechanical) may predispose to back disability. Clinical variables such as pain may affect the patient ability to move and also may result in muscle spasm that led to more pain and movement restriction. Further, functional capabilities may affect the patient and when reduced may lead to disability. Moreover, biomechanical factors such as abnormal posture creates abnormal stress and strain in many spinal structures which are considered predisposing factors for pain and disability.

There is a gab of evidence to examine the relationships between those variables and to predict disability in patients with chronic nonspecific low back pain using various variables.

ELIGIBILITY:
Inclusion Criteria:

- age between 20 and 40 years, either sex, and symptoms lasting longer than three months, which imply chronicity

Exclusion Criteria:

* Pregnancy, Spinal pathologies or surgery, or any other deformities or visual or auditory issues, as well as ongoing physical or medical treatment for LBP

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 100 subjects will be recruited from the university A local advertisement sent via e-mail to the university's postgraduate students and administrative staff
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
back disability using oswestry disability index | 1 month
  oswestry disability index has been designed to give us information as to how your back pain has affected your ability to manage everyday life. For each question, there is a possible 5 points; 0 for the first answer, 1 for the second answer, etc. Add up the total for the 10 questions and rate them on the scale at right.. 0 - 4 No disability 5 - 14 Mild disability 15 - 24 Moderate disability 25 - 34 Severe disability 35 - 50 Completely disabled
back pain intensity using visual analogue scale | 1 month
  visual analogue scale (VAS) is one of the pain rating scales used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
back functional ability using back performance scale | 1 month
  Back performance scale (BPS) has been found to reflect important aspects of physical functioning. It consists of Sock Test, the Pick-up Test, the Roll-up Test, the Fingertip-to-Floor Test, and the Lift Test. For each test a score of 0 was considered a good performance with no signs of activity limitation, a score of 1 was considered a somewhat limited performance, a score of 2 was considered a rather distinct limitation of performance, and a score of 3 was considered a substantially limited performance, if performed at all. The BPS sum score is calculated by adding the individual scores of the 5 tests ranging from 0 to 15.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa M Elabd, Principal Investigator — Benha University
Locations (1):
- Benha University, Cairo, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be available up on reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: up on completion